CLINICAL TRIAL: NCT01303718
Title: INcrease Of VAgal TonE in CHF (INOVATE-HF) - A Randomized Study to Establish the Safety and Efficacy of CardioFit® for the Treatment of Subjects With Heart Failure and Left Ventricular Dysfunction
Brief Title: INcrease Of VAgal TonE in CHF
Acronym: INOVATE-HF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility of Primary Efficacy Endpoint
Sponsor: BioControl Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-05-026
Record Dates: First submitted 2011-02-18; First posted 2011-02-25 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Left Ventricular Dysfunction; Heart Failure
Keywords: LV Dysfunction; Heart Failure
MeSH Terms: conditions — Ventricular Dysfunction, Left; Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CardioFit® System (Experimental): Vagal nerve stimulation with the CardioFit® system
  Interventions: Device: CardioFit® System
- Standard of Care (Active Comparator): Usual care (no CardioFit System implant)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: CardioFit® System — Vagal nerve stimulation with the CardioFit® system
  Arms: CardioFit® System
Other: Standard of Care — Usual care for LV dysfunction and heart failure (no CardioFit System implant)
  Arms: Standard of Care

SUMMARY:
The purpose of the INOVATE-HF study is to demonstrate the long-term safety and efficacy of vagus nerve stimulation with the CardioFit® system for the treatment of subjects with Heart Failure.

DETAILED DESCRIPTION:
Prospective, Randomized (3:2 active:control), Open Label, Event-driven Interventional Study. All subjects undergo the following: Baseline, Randomization, (Implantation & Optimization for subjects randomized to the active therapy), and Follow-up Period, followed by an Extension period, which lasts until the end of the study. The Clinical Events Committee (CEC) and Data Monitoring and Safety Board (DSMB) will conduct scheduled independent reviews of the data at the following time-points in order to ensure that an ongoing acceptable safety profile is being achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic symptomatic heart failure in New York Heart Association functional class III.
2. Age of at least 18 years.
3. Subjects should be predominately in sinus rhythm at the time of enrollment.
4. On stable optimally uptitrated medical therapy recommended according to current guidelines as standard of care for heart failure therapy.
5. LVEF ≤ 40% per site measurement within three months before enrollment.
6. The left ventricular end diastolic diameter, per site measurement, should be between 50 and 80 mm.
7. The subject is a male or postmenopausal female. Females of childbearing age may be included if an acceptable contraception measure is used.
8. Subject must sign an approved informed consent form. Subject agrees to attend all followup evaluations.
9. Subjects with CRT devices may be included in the trial provided they have had CRT for at least 12 months.

Exclusion Criteria:

1. Presence of a life threatening condition or disease other than heart failure, that is likely to lead to death within 6 months.
2. Acute myocardial infarction (MI), variant angina pectoris, unstable angina or acute coronary syndrome in the previous one month.
3. History of stroke or TIA within the previous 3 months or significant neurological damage that would impair the ability to respond to or detect improvement with the vagal nerve stimulation.
4. Coronary Artery Bypass Surgery (CABG), valve replacement or repair, aortic surgery or PCI) in the prior 3 months or planned/anticipated within 6 months.
5. Heart failure due to acute myocarditis, restrictive cardiomyopathy, constrictive pericarditis or hemodynamically significant aortic valve insufficiency, aortic stenosis, or mitral valve stenosis.
6. Severe renal failure (creatinine level > 3 mg/dL (265 micromole/liter).
7. Severe hepatic failure (transaminase level four times ULN, or total bilirubin level > 1.8 mmol/dL).
8. Uncontrolled Diabetes Mellitus, which in the opinion of the investigator, would compromise the safety of the implant procedure and/or the ability to respond or detect improvement with vagal nerve stimulation.
9. Previous right neck surgery, including for cerebrovascular disease (CVD), malignancy, and previous irradiation therapy of the neck, which in the opinion of the implanting surgeon, would preclude safe implantation of the vagal nerve cuff. Subjects with more than 70% right carotid artery stenosis assessed on carotid ultrasound are excluded.
10. Current hypotension (systolic blood pressure below 80 mmHg).
11. Active peptic ulcer disease or history of upper GI bleeding, or ulcer within 6 months.
12. History of lung disease such as severe asthma, COPD (e.g., FEV1<1.5 liter) or continuous oxygen dependence.
13. 2nd or 3rd degree AV block or other pacemaker indication that is not treated with a pacemaker.
14. Chronic atrial fibrillation or flutter in the previous 3 months, or hospitalization for AF due to clinical manifestations of such in the last 6 months.
15. Use of unipolar sensing
16. Congenital or acquired long QT syndrome.
17. Documented recorded or suspected vaso-vagal syncope or vaso depressor syncope.
18. Treatment by investigational drug or device within the past 3 months.
19. The subject must not have received inotropic therapy within 2 months or be considered a possible candidate for inotropic therapy within the next 1 month.
20. Inability to understand the informed consent and/or prior diagnosis of major affective disorder e.g., major depression or bipolar disorder or schizophrenia that requires ongoing treatment and is not adequately controlled by medication.
21. Subjects transplanted with heart or other tissues or organs, or on a heart transplant waiting list and anticipated to receive a transplant within 6 months of randomization.
22. Immunosuppressed subjects; subjects under systemic steroid treatment.
23. Anemia with Hgb ≤ 9.5 g/L. Treatment with erythropoietin or other similar agents is allowed if used to keep Hgb > 9.5 g/L.
24. Untreated obstructive sleep apnea ("OSA") with apnea-hypopnea index of 15 or more; or OSA that is treated for less than 3-months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2011-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants reaching all-cause mortality or unplanned heart failure hospitalization or equivalent. | Until the end of the study
  The primary efficacy end-point of the study is the composite of all-cause mortality or unplanned heart failure hospitalization equivalent using a time to first event analysis, as compared between the two study arms after a pre-specified number of such events have been accumulated.
Co-Primary Safety Endpoints: a) Freedom from procedure and system related complication events and b) Number of all-cause death cases or complications resulting in hospitalization | a) 90 days and b) Until the end of the study
  The co-primary safety endpoints of the study are the following:
  1. Freedom from procedure and system related complication events through 90 days
  2. Demonstrate time to first event equivalence in all-cause mortality and complications resulting in prolonged hospitalization between the Control and CardioFit

SECONDARY OUTCOMES:
The rate of unplanned heart failure hospitalization equivalents | Until the end of the study
  The rate of unplanned heart failure hospitalization equivalents
Mean improvement in LVESVi from baseline to 12-months | 12 Months
  Mean improvement in LVESVi from baseline to 12-months
Mean improvement in the summary score of the KCCQ from baseline to 12-months | 12 Months
  Mean improvement in the summary score of the KCCQ from baseline to 12-months
Mean improvement in 6 minute walk test from baseline to 12-months | 12 Months
  Mean improvement in 6 minute walk test from baseline to 12-months
All cause mortality and the number of unplanned heart failure hospitalization equivalents | Until the end of the study
  All cause mortality and the number of unplanned heart failure hospitalization equivalents
Rate of hospitalization-free days | Until the end of the study
  Rate of hospitalization-free days
Secondary Safety Endpoints: Mortality and Complications | Until the end of the study
  The following additional (secondary) safety endpoint data will also be evaluated comparatively at 6- and 12-months:
  1. All-cause mortality
  2. Cardiovascular mortality
  3. Serious adverse events
  4. Complications
  5. System- or procedure-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Douglas L. Mann, MD, Study Chair — Washington University School of Medicine; Michael Gold, Study Chair — Medical University of South Carolina
Locations (87):
- United States (57):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Banner Research Institute, Mesa, Arizona
  - Glendale Memorial Hospital, Glendale, California
  - Sutter Memorial Hospital, Sacramento, California
  - Chula Vista Heart Clinic, San Diego, California
  - South Denver Cardiology, Denver, Colorado
  - Clearwater Cardiovascular Consultants/Morton Plant, Clearwater, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Florida Hospital, CV Research Institute, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - St. Joseph's Hospital, Atlanta, Georgia
  - Georgia Arrhythmia Consultants, Macon, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Community Heart and Vascular Clinic, Indianapolis, Indiana
  - Saint Vincent Medical Group, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Detroit Medical Center - Harper Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Detroit Clinical Research Center/Botsford Hospital, Farmington Hills, Michigan
  - Michigan Cardiovascular Institute, Saginaw, Michigan
  - Munson Medical Center/Traverse Heart and Vascular, Traverse, Michigan
  - Park Nicollet / Methodist, Saint Louis Park, Minnesota
  - United Heart & Vascular, Saint Paul, Minnesota
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - St. Luke's Mid America Heart Institute, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Bryan Heart Institute, Lincoln, Nebraska
  - Health Care Partners Cardiology/St. Rose Hospital, Las Vegas, Nevada
  - Mount Sinai, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center/Albert Einstein Colelge of Medicine, The Bronx, New York
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State, Columbus, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Hershey Medical Center/Penn State, Hershey, Pennsylvania
  - Lancaster Heart and Stroke Foundation, Lancaster, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - VA Tennessee Valley Healthcare System, Nashville, Tennessee
  - Lone Star Heart Center, Amarillo, Texas
  - Texas Cardiac Arrhythmia (TCA), Austin, Texas
  - Dallas Cardiovascular Associates (CRSTI), Dallas, Texas
  - EP Heart/ETHSC at Houston, Houston, Texas
  - St Lukes Episcopal, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Sentara Norfolk Hospital, Norfolk, Virginia
  - Kootenai Heart Clinic, Spokane, Washington
  - Multicare Health System, Tacoma, Washington
  - Aurora Health Care, Lake Geneva, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
- Belgium (3):
  - Onze Lieve Vrouwziekenhuis, Aalst
  - Ziekenhuis Oost Limburg, Genk
  - Universitair Ziekenhuis Campus Gasthuisberg, Leuven
- Germany (9):
  - Uniklinikum Aachen, Aachen
  - Charite Benjamin Franklin Campus, Berlin
  - Charite Campus Virchow-Klinikum Medizinische Klinik mit Schwerpunkt Kardiologie, Berlin
  - St. Josef Hospital, Bochum
  - Asklepios St Georg Hospital, Hamburg
  - Albertinen-Krankenhaus, Hamburg
  - MHH Klinik für Kardiologie und Angiologie, Hanover
  - University of Medicine Mannheim, Mannheim
  - Uniklinikum Muenster, Münster
- Bnai-Zion Hospital, Haifa, Israel
- Netherlands (3):
  - University Medical Centre Groningen, Groningen
  - Maastricht University Medical Center, Maastricht
  - Erasmus University Medical Center Rotterdam, Rotterdam
- Poland (2):
  - Fourth Military Hospital Wroclaw, Wroclaw
  - Medical University of Łodź, Łodź
- Serbia (2):
  - Clinical Centre of Serbia, Belgrade
  - Clinical Hosptial Centre Bezanijska Kosa, Belgrade
- United Kingdom (10):
  - Golden Jubilee National Hospital, Clydebank, Scotland
  - Queen Elizabeth Hospital, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - St. Peter's Hospital, Chertsey
  - University of Hull/Castle Hill Hospital, Cottingham
  - University Hospital Coventry, Coventry
  - Glenfield Hospital, Leicester
  - Royal Brompton Hospital, London
  - Oxford University/John Radcliffe Hospital, Oxford
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Gold MR, Van Veldhuisen DJ, Hauptman PJ, Borggrefe M, Kubo SH, Lieberman RA, Milasinovic G, Berman BJ, Djordjevic S, Neelagaru S, Schwartz PJ, Starling RC, Mann DL. Vagus Nerve Stimulation for the Treatment of Heart Failure: The INOVATE-HF Trial. J Am Coll Cardiol. 2016 Jul 12;68(2):149-58. doi: 10.1016/j.jacc.2016.03.525. Epub 2016 Apr 4. PMID 27058909
- [Derived] Hauptman PJ, Schwartz PJ, Gold MR, Borggrefe M, Van Veldhuisen DJ, Starling RC, Mann DL. Rationale and study design of the increase of vagal tone in heart failure study: INOVATE-HF. Am Heart J. 2012 Jun;163(6):954-962.e1. doi: 10.1016/j.ahj.2012.03.021. PMID 22709747
- See also: CardioFit Pilot Study Description and Results — http://clinicaltrials.gov/ct2/show/NCT00461019